CLINICAL TRIAL: NCT02673177
Title: A Randomized, Prospective Trial of Robotic Versus Laparoscopic-assisted Radical Resection for Rectal Cancer in Urinary, Erectile Function and Anal Function
Brief Title: Trial of Robotic Versus Laparoscopic-assisted Radical Resection for Rectal Cancer
Acronym: TRVL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Tang Bo, Principal Investigator, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015(43)
Record Dates: First submitted 2016-01-27; First posted 2016-02-03 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Rectal Neoplasms
Keywords: robot-assisted total mesorectal excision(RTME); laparoscopic total mesorectal excision(LTME); urinary function; sexual function; sphincter- preservation; low rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot-assisted total mesorectal excision (Experimental): Robot-assisted total mesorectal excision (RTME) for rectal cancer. Two different RTME procedures were chose to personalized patients. Generally, when the tumor located within 5-15cm from the anal verge, low anterior resection (LAR) was employed, and tumor located below 5cm, abdominoperineal resection (APR) was applied usually.
  Interventions: Procedure: robot-assisted total mesorectal excision
- Laparoscopic total mesorectal excision (Active Comparator): Traditional laparoscopic total mesorectal excision (LTME) for rectal cancer was performed. The Urinary, sexual function and sphincter- preservation outcomes were evaluated.
  Interventions: Procedure: laparoscopic total mesorectal excision

INTERVENTIONS:
Procedure: robot-assisted total mesorectal excision — The Da Vinci Surgical System may help to protect subtle anatomical structure and provide more functional protection when compared to laparoscopic surgery. This study aimed to compare RTME and laparoscopic total mesorectal excision (LTME) for rectal cancer with regard to Urinary, sexual function and sphincter- preservation outcomes.
  Arms: Robot-assisted total mesorectal excision
Procedure: laparoscopic total mesorectal excision — Traditional laparoscopic total mesorectal excision (LTME) for rectal cancer.
  Arms: Laparoscopic total mesorectal excision

SUMMARY:
This study compared robot-assisted total mesorectal excision (RTME) and laparoscopic total mesorectal excision (LTME) with regard to urinary function, sexual function and sphincter- preservation outcomes for low rectal cancer.

DETAILED DESCRIPTION:
Urinary and sexual dysfunction are recognized complications of rectal cancer surgery in men. This study compared robot-assisted total mesorectal excision (RTME) and laparoscopic total mesorectal excision(LTME) with regard to these functional outcomes.Sphincter- preservation outcomes for low rectal cancer was observed as well.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who are acceptable to two surgical procedures for the robot- assisted or laparoscopy-assisted rectal cancer, are willing to randomized trial;
* 2. Matching the diagnostic criteria;
* 3. Aged 18-70 years old;
* 4. Preoperative TNM staging (CT, laparoscopic exploration): cT1-3N0-3M0 (excluding M1, T4);
* 5. Preoperative ASA 3 scores;
* 6. There was no history of malignancy, no other malignant tumors by preoperative examination;
* 7. Without undergoing definitive treatment, such as radiotherapy, chemotherapy or immunotherapy preoperatively;
* 8. The informed consent form was signed by the patient himself(herself)or his principal agent;
* 9. In accordance with the international erectile function questionnaire (IIEF) urinary function scale, The urinary sexual function are normal.

Exclusion Criteria:

* 1. Age less than 18 years old or more than 70 years old;
* 2. Previous psychiatric patients or patients refused to sign the informed consent;
* 3. Attending other related clinical studies on surgical treatment of rectal cancer;
* 4. The patient has a history of malignant tumor, or a combination of other malignant tumors;
* 5. Patients have been treated with definitive treatment: radiotherapy, chemotherapy or immunotherapy;
* 6. Patients had received otherper abdominal operations (except for laparoscopic cholecystectomy);
* 7. ASA >3;
* 8. Laparoscopic surgical contraindications: such as severe heart lung disease; abdominal wall hernia; diaphragmatic hernia; coagulation disorder; portal hypertension; pregnancy, etc.;
* 9. Those who has been confirmed to be unable to do a radical resection (T4 stage) for local advanced tumor;
* 10. Those who have urination sexual dysfunction preoperatively.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of sexual and urinary dysfunction | One years after surgery

SECONDARY OUTCOMES:
disease-free survival(DFS ) | 3 years disease-free survival
  DFS was defined as from the date of randomization to the date of tumor recurrence or death from any cause
Anus preservation rate | One years after surgery

IPD SHARING:
Plan to Share IPD: Yes